CLINICAL TRIAL: NCT02518269
Title: A Prospective 3-Arm Randomized Controlled Study on G7 Acetabular Cup With Echo BiMetric Stem in Total Hip Arthroplasty
Brief Title: A 3-Arm Study on G7 Acetabular Cup With Echo BiMetric Stem in Total Hip Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTHO.CR.GH33
Record Dates: First submitted 2015-04-29; First posted 2015-08-07 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthrosis; Pain; Arthritis
Keywords: hip; arthroplasty; G7; EchoBimetric; E1; ceramic; Arcom XL
MeSH Terms: conditions — Osteoarthritis; Pain; Arthritis | interventions — Arthroplasty, Replacement, Hip; methyl N-acetylsibirosaminide; Pentosan Sulfuric Polyester

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G7 MoP (Arcom XL) + Echo BiMetric (Active Comparator): Eligible patients will be enrolled and planned for Hip Arthroplasty and operated with the Echo BiMetric femoral stem and G7 Acetabular cup. This group will receive an Arcom Xl liner and a metal head
  Interventions: Procedure: Hip Arthroplasty
- G7 MoP (E1) + Echo BiMetric (Active Comparator): Eligible patients will be enrolled and planned for Hip Arthroplasty and will be operated with the Echo BiMetric femoral stem and G7 Acetabular cup. This group will receive an E1 liner and a metal head.
  Interventions: Procedure: Hip Arthroplasty
- G7 CoC + Echo BiMetric (Active Comparator): Eligible patients will be enrolled and planned for Hip Arthroplasty and operated with the Echo BiMetric femoral stem and G7 Acetabular cup. This group will receive a ceramic liner and a ceramic head
  Interventions: Procedure: Hip Arthroplasty

INTERVENTIONS:
Procedure: Hip Arthroplasty — Hip Arthroplasty comparing 3 different bearings.
  Other Names: G7 acetabular cup system,; Echo Bimetric Full profile stem; Neutral liner, Arcom XL; Neutral liner, E1; Ceramic liner; Monobloc Ceramic Biolox Delta Head, 32 mm; Cobolt chrome head, 32 mm; porous coated (PPS) titanium alloy shells

SUMMARY:
The study is designed to compare three articulation options in terms of osteolysis, patient satisfaction, clinical and radiographic outcomes (Oxford Hip score (OHS) and Harris Hip score (HHS) and safety.

In addition, the purpose of the study is also to evaluate the safety and effectiveness of patients who received G7 Acetabular system in conjunction with Echo BiMetric stem in primary total hip arthroplasty.

DETAILED DESCRIPTION:
DESIGN: Prospective 3 Arm Randomized controlled trial.

PURPOSE:To compare three commonly used contemporary bearings in Total Hip Arthroplasty (THA). In addition, to evaluate the safety and effectiveness of the G7 Cups and Echo BiMetric Stem in THA.

OUTCOME MEASURES: Osteolysis, clinical outcomes, patient satisfaction, intraoperative/surgical data, implant positioning, survivor ship, and adverse events.

POPULATION: 360 hips (240 will have CT scan for analysis of osteolysis).

ELIGIBILITY: Patients who meet inclusion and exclusion criteria defined in this protocol.

DURATION: All patients will be followed at 3 months, 1, 2, 5, 7 and 10 year postoperatively. Assuming the enrollment will be completed 18 months. The total study duration will be 11.5 years.

STUDY GROUPS/TREATMENTS

Group 1 - G7 Metal-on-Polyethylene (MoP) (Arcom XL) + Echo BiMetric Group 2 - G7 Metal-on-Polyethylene (MoP) (E1) + Echo BiMetric Group 3 - G7 Ceramic-on-Ceramic (CoC) + Echo BiMetric The study's primary efficacy endpoint will include the difference in osteolytic volume at 5 years postoperatively measured by Computertomografi (CT) scan.

ELIGIBILITY:
Inclusion Criteria:

Patient is 18 to 75 years of age, inclusive.

* Patients determined to be suitable for uncemented fixation by investigator
* Patient is skeletally mature.
* Patient qualifies for primary unilateral total hip arthroplasty (THA) based on physical exam and medical history including the following:

  * Osteoarthritis (OA)
  * Developmental Dysplasia without subluxation
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.

Exclusion Criteria:

The patient is:

* A prisoner
* Mentally incompetent or unable to understand what participation in the study entails
* A known alcohol or drug abuser
* Anticipated to be non-compliant.

  * The patient has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
  * The patient has a neurologic condition in the ipsilateral or contralateral limb which affects lower limb function.
  * The patient has a diagnosed systemic disease that could affect his/her safety or the study outcome.
  * The patient is known to be pregnant.
  * The patient is unwilling or unable to give informed consent, or to comply with the follow-up program.
  * The patient has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.

The patient has had previous Girdlestone procedure (resection arthroplasty) or surgical fusion of the hip to be operated.

* The patient has insufficient bone stock to fix the component. Insufficient bone stock exists (ex: Dorr type C) in the presence of metabolic bone disease (i.e. osteoporosis), cancer, and radiation.
* Estimated cup size smaller than 48 or stem size smaller than 7
* The patient has known local bone tumors in the operative hip.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Difference in osteolytic volume at 5 years postoperatively measured by CT scan. | 5 years
  CT scan will be performed on 240 of the 360 patients post operatively and at 5 years follow up

SECONDARY OUTCOMES:
Hip specific clinical outcome in patients who received the one of the above mentioned combinations of total hip systems. | 3 months, 1,2,5,7 and 10 year follow up
  Oxford Hip score (OHS) will be collected from all the patients preoperative and at all follow up visits.
Implant positioning | Immediately postoperative,1,2,5,7 and 10 year follow up
  Implant positioning will be measured using Martell method .
Subjective satisfaction | 3 months, 1,2,5,7 and 10 year follow up
  Subjective satisfaction will be collected using Numerical Rating Scale (NRS) and will be collected preoperative and at all follow ups.
Safety and survivorship | Continously throughout the study until 10 years FU
  Adverse Events will be reported including revisions at any post-operative time points
Squeaking evaluation | 3 months, 1,2,5,7,10 years
  Evaluation of noise from the hip will be made at all follow up visits by a noise assessment form
Pain Assessment | 3 months, 1,2,5,7,10 years
  Pain will be collected using Numerical Rating Scale (NRS) and will be collected preoperative and at all follow ups.
Health related quality of life | 3 months, 1,2,5,7,10 years
  EQ5D (Health related quality of life questionnaire from Euro Qol) will be collected from all the patients preoperative and at all follow up visits.
Physical activity level | 3 months, 1,2,5,7,10 years
  UCLA (University California Los Angeles activity questionnaire) will be collected from all the patients preoperative and at all follow up visits.
Hip specific clinical patient outcome measure | 3 months, 1,2,5,7,10 years
  Harris Hip score (HHS)will be collected from all the patients preoperative and at all follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, MD, PhD, Principal Investigator — Hvidovre University Hospital; Henrik Malchau, MD, PhD, Principal Investigator — Sahlgrenska University Hospital; Ville Remes, MD, PhD, Principal Investigator — Jokilaakson Terveys Oy
Locations (5):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Hvidovre hospital, Copenhagen
- Finland (2):
  - Jokilaakson Terveys Oy, Jämsä
  - Turku university hospital, Turku
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Plan is to publish articles for all the enrolled patients.